CLINICAL TRIAL: NCT02071121
Title: A Randomized, Double-Blinded, Placebo-Controlled, Single-Ascending-Dose (SAD) Study of the Safety, Tolerability, and Pharmacokinetics of BIIB061 in Healthy Adult Volunteers Including Absolute Bioavailability and Food Effect
Brief Title: Single Ascending Dose Study of the Safety, Tolerability, and Pharmacokinetics of BIIB061 in Healthy Adult Volunteers Including Absolute Bioavailability and Food Effect
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 231HV101
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
Keywords: BIIB061; Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo (Placebo Comparator): Fasted participants will receive a single oral dose of placebo to BIIB061.
  Interventions: Drug: Placebo
- BIIB061 3 mg (Experimental): Fasted participants will receive a single oral dose of BIIB061 3 mg.
  Interventions: Drug: BIIB061
- BIIB061 10 mg (Experimental): Fasted participants will receive a single oral dose of BIIB061 10 mg followed by a tracer amount of 14C-BIIB061 (at ≤ 500 nCi/participant; approximately 4 μg of BIIB061), administered by manual slow intravenous push injection at 4 hours postdose.
  Interventions: Drug: BIIB061; Drug: 14C-BIIB061
- BIIB061 30 mg (Experimental): Fasted participants will receive a single oral dose of BIIB061 30 mg. Following a washout period, participants will receive the same dose of BIIB061 after a high-fat, high-calorie meal (fed state).
  Interventions: Drug: BIIB061
- BIIB061 60 mg (Experimental): Fasted participants will receive a single oral dose of BIIB061 60 mg.
  Interventions: Drug: BIIB061
- BIIB061 100 mg (Experimental): Fasted participants will receive a single oral dose of BIIB061 100 mg.
  Interventions: Drug: BIIB061

INTERVENTIONS:
Drug: BIIB061 — BIIB061 capsules for oral administration
  Arms: BIIB061 10 mg; BIIB061 100 mg; BIIB061 3 mg; BIIB061 30 mg; BIIB061 60 mg
Drug: Placebo — BIIB061 matching placebo capsules
  Arms: Placebo
Drug: 14C-BIIB061 — Radiolabeled containing 14C-BIIB061 ≤ 500 nCi.
  Arms: BIIB061 10 mg

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of single doses of BIIB061 administered to healthy adult volunteers. Secondary objectives in this study population are to determine the single-dose pharmacokinetic (PK) profile and the absolute bioavailability (Fabs) of BIIB061 and to determine the effects of food intake (high-fat, high-calorie meal) on BIIB061 PK and safety.

ELIGIBILITY:
Key Inclusion Criteria:

* Males and postmenopausal (defined as no menses for 12 months and confirmed by follicle-stimulating hormone (FSH) levels determined at screening to be in the postmenopausal range) or surgically sterile females.
* All males must practice effective contraception during the study and be willing and able to continue male contraception for 3 months after the dose of study treatment. All male participants must also be willing to refrain from sperm donation for at least 3 months after their last dose of study treatment. Note: Females of childbearing potential, are not allowed to enter the study.
* Must be in good health and have normal vital signs as determined by the Investigator.
* Participants agree to abstain from alcohol ingestion for the duration of time that they are in the study.
* Must be a nonsmoker and must not use chewing tobacco or nicotine products, for at least 3 months prior to Day -1.
* Must have a body mass index (BMI) of 18 to 30 kg/m2, inclusive.

Key Exclusion Criteria:

* History of or positive test result at screening for human immunodeficiency virus (HIV).
* History of any clinically significant cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, oncologic, or other major disease, as determined by the Investigator.
* Clinically significant (as determined by the Investigator) 12-lead electrocardiogram (ECG) abnormalities, including corrected QT interval using Fridericia's correction method of >450 ms for males and >470 ms for females.
* History of severe allergic or anaphylactic reactions.
* Serious infection (e.g., pneumonia, septicemia) as determined by the Investigator, within 3 months prior to Day -1.
* Consumption of grapefruit or grapefruit-containing products within 3 days of dosing.
* Treatment with any over-the-counter products, including herbal and/or alternative health preparations and procedures within the 14 days prior to Day -1.
* Current enrollment in any other drug, biologic, device, or clinical study, or treatment with an investigational drug or approved therapy for investigational use within 30 days (or 5 half-lives, whichever is longer) prior to Day -1.
* Blood donation (1 unit or more) within 30 days prior to Day -1
* History of drug or alcohol abuse (as determined by the Investigator), a positive urine drug/alcohol test, or a positive cotinine test at Screening or Day -1, or alcohol use within 48 hours (as reported by the subject) prior to Day -1.
* Vigorous exercise (as determined by the Investigator) within 48 hours prior to Day -1.
* History of malignant disease, including solid tumors and hematologic malignancies.
* Surgery within 3 months prior to Day-1.
* History of seizures other than childhood febrile seizure.
* Inability or unwillingness to comply with study requirements.

NOTE: Other protocol-defined inclusion/exclusion criteria may apply

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2013-12; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Number of participants that experience adverse events (AEs) and Serious Adverse Events (SAEs) | 28 days

SECONDARY OUTCOMES:
Area under the concentration-time curve from time 0 to infinity (AUCinf) of BIIB061 | Predose and up to 28 days post-dose.
Maximum observed concentration (Cmax) of BIIB061 | Predose and up to 28 days post-dose.
Time to reach maximum observed concentration (Tmax) of BIIB061 | Predose and up to 28 days post-dose.
Half-life (t1/2) of BIIB061 | Predose and up to 28 days post-dose.
Absolute bioavailability (Fabs) of BIIB061 for the absolute bioavailability cohort only | Predose and up to 28 days post-dose.
Clearance of BIIB061 for the absolute bioavailability cohort only. | Predose and up to 28 days post-dose.
Volume of distribution (Vd) of BIIB061 for the absolute bioavailability cohort only. | Predose and up to 28 days post-dose.
The difference between PK parameters (AUC, Cmax, Tmax, and t1/2) taken under fasting conditions and following a high-fat, high-calorie meal are analyzed | Day 1 to Week 4 (28-day fasting PK measurements), a washout period followed by dosing after a high-fat, high-calorie meal (28-day PK measurements)
  For the fasting PK portion of the study, participants' PK samples are taken after an overnight fast of at least 10 hours. For the food effect portion of the study, the dose is given 30 minutes following a high-fat, high-calorie meal.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (2):
- United States (2):
  - Research Site, Evansville, Indiana
  - Research Site, Madison, Wisconsin